CLINICAL TRIAL: NCT03129841
Title: Effects of Late Dinner Against Early Dinner on Weight Loss Healthy Obese Women in a Weight-loss Program: a Randomized Clinical Trial
Brief Title: Effects of Late Dinner Against Early Dinner on Weight Loss Healthy Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novindiet Clinic (Other)
Collaborators: University of Nottingham (Other); Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ND-202
Record Dates: First submitted 2017-04-15; First posted 2017-04-26 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Obesity; Overweight
Keywords: weight loss; dietary pattern; late dinner; early dinner
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early dinner+Diet (Experimental)
  Interventions: Behavioral: Early dinner+Diet
- late dinner+Diet (Experimental)
  Interventions: Behavioral: Late dinner+Diet

INTERVENTIONS:
Behavioral: Early dinner+Diet — Subjects are asked to eat dinner meals between 7:00- 7:30 PM in the ED group, while they are on a multidisciplinary weight loss plan for 12 weeks.
  Other Names: ED
  Arms: early dinner+Diet
Behavioral: Late dinner+Diet — Subjects are asked to eat their dinner meal between 10:30-11:00PM, while they are on a multidisciplinary weight loss plan for 12 weeks.
  Other Names: LD
  Arms: late dinner+Diet

SUMMARY:
The aim of the present study is to test whether late eating dinner could affect the amount of weight loss in healthy obese women in a weight-loss program.

ELIGIBILITY:
Inclusion Criteria:

* Must have Body mass index (BMI) between 27-35 kg/ m².
* Must be able to have moderate exercise.
* Must be interested to have weight loss.

Exclusion Criteria:

* Participating in a research project involving weight loss or physical activity in the previous six months.
* Pregnancy or lactation during the previous 6 months, or planned pregnancy in the next six months.
* Taking medication that could affect metabolism or change body weight.
* Report heart problems, chest pain, and cancer within the last five years.
* Smoking
* Menopause
* Diagnosis of any chronic disease such as fatty liver, cancer, chemo/radio therapy, heart disease, immune compromised conditions, abnormal thyroid hormone level.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-11-18 (Actual)

PRIMARY OUTCOMES:
weight loss | 12 Weeks
  kg

SECONDARY OUTCOMES:
waist circumference | 12 Weeks
  cm
fasting plasma glucose | 12 Weeks
  mmol/L
insulin level | 12 Weeks
  mU/l
insulin resistance (HOMA-IR) | 12 Weeks
  Score
glycosylated hemoglobin (HbA1c) | 12 Weeks
  percentage (%)
lipid profiles | 12 Weeks
  mmol/l
Liver Enzyme (SGOT, SGPT) | 12 Weeks
  U/l

CONTACTS AND LOCATIONS:
Locations (1):
- NovinDiet Clinic, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided